CLINICAL TRIAL: NCT02054416
Title: External Compression Therapy for Secondary Prevention of Lower-Limb Loss and Cardiovascular Mortality in Underserved Philadelphia Patient Population: A Randomized Controlled Study
Brief Title: External Compression Therapy for Secondary Prevention of Lower-Limb Loss and Cardiovascular Mortality
Acronym: ArtAssist
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PVB012013
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-10

CONDITIONS: Critical Limb Ischemia
Keywords: non-traumatic lower limb amputation; AKA; BKA
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Art Assist Device (Active Comparator): The ArtAssist© (model AA1000) device is made by ACI Medical located in San Marcos, CA (http://acimedical.com/) and is cleared per FDA under K942530.The study intervention will consist of one hour of IPC with the ArtAssist© device to the remaining leg, three times a day for a three month period. We will obtain the usage data from the device when the subject returns the device (the device has an internal device that stores the usage data) to evaluate subject compliance.
  Interventions: Device: ArtAssist© Device
- Sham Device (Sham Comparator): Sham devices look identical to the actual ArtAssist© devices, but provide low-pressure and differ only in number-coded tubing. The study "sham intervention" will consist of one hour of IPC with the sham ArtAssist© device to the remaining leg, three times a day for a three month period. We will obtain the usage data from the device when the subject returns the device (the sham device has an internal device that stores the usage data) to evaluate subject compliance.
  Interventions: Device: ArtAssist© Device

INTERVENTIONS:
Device: ArtAssist© Device — The study intervention will consist of one hour of IPC with the ArtAssist© device to the remaining leg, three times a day for a three month period. We will obtain the usage data from the device when the subject returns the device (the device has an internal device that stores the usage data) to evaluate subject compliance.
  Other Names: The ArtAssist© (model AA1000)

SUMMARY:
In this clinical research study the investigators will test the efficacy of an innovative, non-invasive methodology to reduce mortality and lower limb loss among high-risk medically-underserved patients with cardiovascular disease in North Philadelphia.

Patients with cardiovascular disease and recent lower limb amputation will be treated with an intermittent compression device on the remaining lower limb to prevent dual amputation.

The study hypothesis is that the study intervention will protect against further lower limb-loss/death and reduce cardiovascular mortality in these patients (one year effect against limb-loss/death).

This study may result in better secondary prevention strategies for disadvantaged urban populations as well as the general population.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate whether a non-invasive intervention for 3 months with an intermittent compression device (ArtAssist®) in a high risk patient group reduces the risk of subsequent one-year limb-loss and/or death (e.g. one-year amputation-free survival and overall survival.) Survival after an amputation is markedly decreased due to generalized cardiovascular disease. The thirty-day mortality after amputation ranges from 6% to 16% depending on renal function. Two-year mortality after amputation is up to 40%.For dialysis patients, two year mortality was 58%.13 The five-year mortality after amputation in non-renal patients is 65%, while in dialysis patients five-year mortality is 83%. Patients who have undergone a major lower extremity amputation related to vascular disease are also at increased risk for losing their remaining lower extremity. The loss of the second lower extremity has a more profound impact on patients' ability to ambulate or function independently than the first amputation. Despite intensive initial rehabilitation, the use of prosthetics in bilateral amputees decreases rapidly over time. Contra-lateral amputations occur in up to 33%, after a mean of eight months. According to another study, 17% of diabetic initial amputees become bilateral amputees after a median time of less than one year for men and less than two years for women. According to a 2013 study, the majority of the subsequent contra-lateral amputations occur in the first year after the index amputation.

We hope to prove that that there is a role for IPC in vascular patients at high-risk for mortality and limb-loss with relatively low-cost compression therapy. We hope to learn more about which underserved patient categories are most likely to benefit from this and when to start the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female ages ≥ 21years old
* Able and willing to provide informed consent
* Status post amputation of lower limb
* IPC treatment can be initiated within 30 days post lower limb amputation
* Ankle-brachial index in the remaining extremity of less than 0.80, or toe- brachial index less than 0 .60 (obtained within last 6 months)
* Patients must be able to sit and able to perform the compression therapy independently
* Intact renal function or if patient has chronic kidney disease a pre study Creatinine will be obtained. If the patient has acute renal failure or is a dialysis patient he/she is eligible, but will be separately randomized and analyzed because Creatinine is linked to survival.

  * Subjects status post healed minor (toe/metatarsal) amputations on treatment leg will be included.

Exclusion Criteria:

* Patients who have no demonstrable peripheral artery disease by ankle-pressure and/or toe-pressure in the remaining limb (initial amputations were mostly precipitated by diabetic neuropathy, deformity, infection, or acute embolization. Amputations resulting from the late effects of trauma, burns, frostbite, etc. are also excluded.
* Patients who are not able to consent due to their mental status, or who are not willing or able to perform the compression therapy in a sitting position
* Contracted nursing-home patients with index amputations resulting from largely pressure-related tissue-loss decubitus
* Patients with infected gangrene or osteomyelitis present in the contra-lateral extremity (which would need to be compressed) at the time of the index amputation
* Patients with active dry gangrene on the leg that is to be compressed
* Patients with congestive heart failure
* Patients in which a deep venous thrombosis or pulmonary embolism is suspected
* Patients who have undergone arterial compression therapy within 1 year prior to study
* Bilateral amputation of lower extremity
* Patients with an expected life-span less than 3 months
* Patients who require intensive care are not eligible, until they can be transferred to a regular nursing floor
* Patients in whom the remaining limb is non-functional, for example due to previous stroke

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-10; Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Amputation free survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Paul van Bemmelen, MD, PhD, Principal Investigator — Temple University
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States